CLINICAL TRIAL: NCT04063046
Title: Effect of Anesthesia Technique on Early Outcome in Diabetic Patients Undergoing Lower Extremity Amputation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2019-0613
Record Dates: First submitted 2019-08-16; First posted 2019-08-21 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Anesthesia, General

STUDY DESIGN:
Intervention Model Description: A Randomized, outcome assessor-Blinded, Trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Active Comparator): General anesthesia involving intubation or supraglottic airway device insertion
  Interventions: Drug: General anesthesia
- peripheral nerve block (Experimental): popliteal sciatic nerve block
  Interventions: Drug: Peripheral nerve block

INTERVENTIONS:
Drug: General anesthesia — General anesthesia is induced with propofol (0.5-2mg / kg), remifentanil (4-8㎍ / kg / hr) and rocuronium (0.4 ~ 0.6 mg / kg) involving laryngeal mask(supraglottic airway device) insertion or endotracheal intubation. Anesthesia is maintained with 1.0-2.5% sevoflurane and remifentanil.
  Arms: General anesthesia
Drug: Peripheral nerve block — ultrasound-guided popliteal sciatic nerve block is performed
  Arms: peripheral nerve block

SUMMARY:
The aim of this study was to compare

1. early prognosis (mortality, morbidity)
2. changes in concentrations of serum syndecan-1,partial pressure of oxygen(on arterial blood gas analysis), perioperative transfusion, intraoperative vasopressor use between general anesthesia and nerve block in diabetic patients undergoing limb amputation surgery as a prospective randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients undergoing diabetic foot limb amputation.
* 2. Patients aged 20 or older and who meet American Society of Anesthesiologists (ASA) physical class 3-4

Exclusion Criteria:

* 1. patients with dementia or cognitive impairment
* 2. Patients who had previously undergone diabetic foot limb amputation within 1 month.
* 3. If the subject includes a person who can not read the written consent (eg, illiterate, foreigner, etc.)
* 4. pregnant or lactating women
* 5. Contraindications to nerve block (infection of the injection site, no cooperation, patient rejection, history of allergy ro local anesthetics)
* 6. Relative contraindications to general anesthesia (if difficult airways are expected, history of malignant hyperthermia, moderate or severe asthma)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
early prognosis (mortality) | 30days after surgery
  death within 30days after surgery
early prognosis (Unexpected return To The Operation Room) | 30days after surgery
  Indicate whether the patient was unexpectedly returned to the Operation Room during this hospital visit.
early prognosis (Renal failure) | 30days after surgery
  Indicate whether the patient had acute renal failure or worsening renal function resulting in ONE OR BOTH of the following:
  1. Increase in serum creatinine level 3.0 x greater than baseline, or serum creatinine level >=4 mg/dL. Acute rise must be at least 0.5 mg/dl
  2. A new requirement for dialysis postoperatively.
early prognosis (Pneumonia) | 30days after surgery
  Indicate if the patient experienced pneumonia in the postoperative period. Pneumonia is defined as meeting three of five characteristics: fever, leucocytosis, CXR with infiltrate, positive culture from sputum, or treatment with antibiotics.
early prognosis (Respiratory failure) | 30days after surgery
  Indicate whether the patient experienced respiratory failure in the postoperative period requiring mechanical ventilation and/or reintubation.
early prognosis (DVT Requiring Treatment) | 30days after surgery
  Indicate whether the patient has experienced a deep venous thrombosis (DVT) confirmed by doppler study, contrast study, or other study that required treatment.
early prognosis (Myocardial Infarct) | 30days after surgery
  Indicate if the patient experienced a MI postoperatively as evidenced by:
  1. Transmural infarction: Defined by the appearance of a new Q wave in two or more contiguous leads on ECG, or
  2. Subendocardial infarction: (non-Q wave) Infarction, which is considered present in a patient having clinical, angiographic, electrocardiographic, and/or
  3. Laboratory biomarker (CPK,Troponin) evidence of myocardial necrosis with an ECG showing no new Q waves
early prognosis (Surgical Site Infection) | 30days after surgery
  Indicate the extent of surgical site infection if one was present within 30 days of surgery.
early prognosis (New Central Neurological Event) | 30days after surgery
  Indicate whether the patient experienced any of the following neurological events in the postoperative period that was not present preoperatively:
  1. A central neurologic deficit persisting postoperatively for > 72 hours.
  2. A postoperatively transient neurologic deficit (TIA recovery within 24 hours; RIND recovery within 72 hours).
  3. New postoperative coma that persists for at least 24 hours secondary to anoxic/ischemic and/or metabolic encephalopathy, thromboembolic event or cerebral bleed.
early prognosis (Delirium) | 30days after surgery
  Indicate whether the patient experienced delirium in the postoperative period marked by illusions, confusion, cerebral excitement, and having a comparatively short course.

SECONDARY OUTCOMES:
changes in concentrations of serum syndecan-1 | within 5 minutes before start of anesthesia(anesthetic drug injection)
changes in partial pressure of oxygen by arterial blood gas analysis | within 5 minutes before start of anesthesia(anesthetic drug injection)
changes in concentrations of serum syndecan-1 | 1 hour after end of operation
changes in partial pressure of oxygen by arterial blood gas analysis | 1 hour after end of operation
perioperative transfusion | Intraoperation
perioperative transfusion | Postoperative 48hours
intraoperative vasopressor use | Intraoperation

CONTACTS AND LOCATIONS:
Overall Officials: Yong Seon Choi, Principal Investigator — Severance Hospital
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea